CLINICAL TRIAL: NCT04950699
Title: Peking University and University of Michigan- Study of Myocardial Infarction and Atherosclerosis
Brief Title: Peking University & University of Michigan Study of MI and Atherosclerosis
Acronym: PUUMA
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Peking University First Hospital (Other); Wuhan Asia Heart Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2012092
Record Dates: First submitted 2021-06-27; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Coronary Heart Disease
Keywords: Single-nucleotide Polymorphism; Dyslipidemia
MeSH Terms: conditions — Coronary Disease; Dyslipidemias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Patients without typical symptoms of coronary heart disease, and coronary angiography or coronary CT showed no significant stenosis (coronary stenosis less than 30%), they were non coronary heart disease group, namely control group.
  Interventions: Genetic: Single-nucleotide Polymorphism of genes related with Dyslipidemia
- myocardial infarction: This group includes acute myocardial infarction (ST segment elevation and non ST segment elevation) and old myocardial infarction. The diagnostic basis of acute myocardial infarction: cardiac biomarkers (cardiac troponin and / or myocardial enzymes) increased or decreased, at least once the value exceeded the upper limit of normal, and there was the following evidence of myocardial ischemia: (1) clinical symptoms of myocardial ischemia（ 2) New changes of myocardial ischemia appeared in ECG, i.e. new ST segment changes or left bundle branch block（ 3) Pathological Q wave appeared in ECG（ 4) Imaging evidence showed new loss of myocardial viability or regional wall motion abnormalities. Diagnosis of old myocardial infarction: the patient provided a history of previous myocardial infarction and confirmed as old myocardial infarction by the third or First Hospital of Peking University.
  Interventions: Genetic: Single-nucleotide Polymorphism of genes related with Dyslipidemia

INTERVENTIONS:
Genetic: Single-nucleotide Polymorphism of genes related with Dyslipidemia — This study is an observational study to study the effect of different genotypes on the incidence of myocardial infarction

SUMMARY:
Coronary heart disease and myocardial infarction have become a major threat to the health of our people. Their incidence rate and mortality rate are still rising. Dyslipidemia is one of the important risk factors. However, little is known about the genetic information of myocardial infarction and dyslipidemia, especially in Chinese population. This project aims to identify new loci related to myocardial infarction and blood lipid level in Chinese population, compare these gene variations with 94 gene variations related to myocardial infarction and blood lipid level in European population, and extract gene variations related to myocardial infarction and blood lipid level in Chinese population. In this case-control study, 3998 blood samples and 702 new blood samples were collected from the sample bank of Peking University Third Hospital and first hospital, respectively. The blood samples were collected from Asian heart disease hospital, Taiyuan cardiovascular disease hospital, Beijing Third Hospital and Shijingshan community follow-up population According to the results of carotid ultrasound or treadmill exercise test, the samples were divided into myocardial infarction group and control group, and the corresponding blood lipid levels were collected. The samples were genotyped by the metabochip gene chip of Illumina company. The data were processed by the calling algorithm of BeadStudio Gentrain 1.0 and the GenoSNP software. The related genes of myocardial infarction were analyzed by logistic regression, and the related genes of blood lipid level were analyzed by linear regression.

DETAILED DESCRIPTION:
Background: coronary heart disease and myocardial infarction have become a major disease threatening the health of our people. Their incidence rate and mortality rate are still rising. Dyslipidemia is one of the important risk factors. However, little is known about the genetic information of myocardial infarction and dyslipidemia, especially in Chinese population.

Objective: to identify new loci related to myocardial infarction and blood lipid level in Chinese population, compare these gene variations with 94 gene variations related to myocardial infarction and blood lipid level in European population, and extract gene variations related to myocardial infarction and blood lipid level in Chinese population.

Methods: This is a case-control study. 9498 blood samples and 702 new blood samples were collected from the sample bank of Peking University Third Hospital and first hospital respectively. The blood samples were collected from Asian heart disease hospital, Beijing Third Hospital and Shijingshan community follow-up population According to the results of carotid ultrasound or treadmill exercise test, the samples were divided into myocardial infarction group and control group, and the corresponding blood lipid levels were collected. The samples were genotyped by the metabochip gene chip of Illumina company. The data were processed by the calling algorithm of BeadStudio Gentrain 1.0 and the GenoSNP software. The related genes of myocardial infarction were analyzed by logistic regression, and the related genes of blood lipid level were analyzed by linear regression.

ELIGIBILITY:
Inclusion Criteria:

- Myocardial infarction group: case group

This group includes acute myocardial infarction (ST segment elevation and non ST segment elevation) and old myocardial infarction. The diagnostic basis of acute myocardial infarction: cardiac biomarkers (cardiac troponin and / or myocardial enzymes) increased or decreased, at least once the value exceeded the upper limit of normal, and there was the following evidence of myocardial ischemia: (1) clinical symptoms of myocardial ischemia（ 2) New changes of myocardial ischemia appeared in ECG, i.e. new ST segment changes or left bundle branch block（ 3) Pathological Q wave appeared in ECG（ 4) Imaging evidence showed new loss of myocardial viability or regional wall motion abnormalities. Diagnosis basis of old myocardial infarction: Patients with previous history of myocardial infarction and confirmed by Peking University Third Hospital, first hospital, Asian heart hospital and Taiyuan cardiovascular hospital.

3.4.2 non coronary heart disease group: control group

The patients in the control group can be enrolled if they meet any of the following criteria: (1) if the patients have no typical symptoms of coronary heart disease, and there is no obvious stenosis on coronary angiography and / or coronary CT (the degree of stenosis in the main coronary artery is less than 30%)（ 2) if the patient had no typical symptoms of coronary heart disease, and the risk factors of coronary heart disease (smoking, hypertension, diabetes, hyperlipidemia, family history of premature coronary heart disease) were not more than 2, no plaque and / or treadmill exercise test were negative for carotid artery ultrasound.

Exclusion Criteria:

* (1) There was severe hepatic and renal insufficiency (2) Cancer and malignant disease patients (3) Severe acute infection or metabolic disorder (4) Acute attack of chronic heart failure (5) Acute myocardial infarction without revascularization within 2 weeks (6) Secondary to obvious valvular heart disease, hypertrophic obstructive heart disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The samples of this study are from Peking University Third Hospital, Peking University First Hospital and Wuhan Asian Heart Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 4700 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
myocardial infarction | Retrospective analysis of cases in 6 years before the start of the study
  This study is a retrospective study, selected patients with myocardial infarction and control group as the research object, no other research endpoint was set

CONTACTS AND LOCATIONS:
Overall Officials: Wei Gao, Dr., Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No